CLINICAL TRIAL: NCT05824000
Title: An Interventional, Non-comparative, Single-center Post Marketing Clinical Follow-up (PMCF) Study to Evaluate Performance and Safety of "Optrex Double Action Soothing and Lubricating Drops"
Brief Title: PMCF Study to Evaluate Performance and Safety of "Optrex Double Action Soothing and Lubricating Drops"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.C. Farmaceutici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COC-R6-CBM
Record Dates: First submitted 2023-04-11; First posted 2023-04-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Allergic Conjunctivitis; Dry Eye; Dry Eye Disease
MeSH Terms: conditions — Conjunctivitis, Allergic; Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyedrops treatment arm (Experimental)
  Interventions: Device: Eye drops for itchy and water eyes

INTERVENTIONS:
Device: Eye drops for itchy and water eyes — Ocular drops for itchy and watery eyes

SUMMARY:
Allergic conjunctivitis (or ocular allergy) and dry eye disease (DED) are two major ocular surface disorders affecting millions of people. A typical clinical symptom of allergic conjunctivitis is itching which is also observed in subjects suffering from DED. Common symptoms of DED also include a foreign body sensation, dryness, irritation, burning sensation and visual disturbance. Patients with allergic conjunctivitis or moderate-to-severe DED may experience a reduced quality of life due to ocular pain, difficulty in performing daily activities, and depression.

Gel-based artificial tear supplements may offer longer retention times and act as a supplement to the mucin layer. Carbomer (also known as Carbopol polymers) is awater-soluble polymeric resin that exhibit excellent viscoelastic and mucoadhesive properties when compared with other polymers. Carbomer is used in liquid or semisolid pharmaceutical, cosmetics, and ophthalmic formulations as rheology modifiers. Aqueous carbomer gels have been used for the treatment of dry eye and allergic conjunctivitis as they provide prolonged ocular residence time of conventional ophthalmic solutions. Furthermore, carbomer has shown compatibility with many active ingredients, good thermal stability, excellent organoleptic characteristics, and good patient acceptance.

For these reasons, an interventional, non-comparative, single-center Post Marketing Clinical Follow-up (PMCF) study was planned to evaluate the performance and safety of "Optrex Double Action soothing and lubricating drops" for itchy and watery eyes.

The objectives of the PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with the use of "Optrex Double Action soothing and lubricating drops" according to the Instructions for Use (IFU).

Each subject, after signing the Informed Consent Form, will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit, "Optrex Double Action soothing and lubricating drops" will be prescribed to the enrolled subject.

The patient will perform 2 on-site visits: V0 and V2/EOS. To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed;
* Male and Female Aged ≥ 18 years at the time of the signature of the ICF;
* Patients with ocular conditions typically associated with itchy and watery eyes (e.g. allergic conjunctivitis, dry eye disease);
* Willing not to use other eye drops during the entire treatment period.

Exclusion Criteria:

* Other - different - eyes clinical conditions (e.g. glaucoma);
* Suspected alcohol or drug abuse.
* Known hypersensitivity or allergy to Investigational Product (IP) components;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. rheumatic disease, diabetes);
* Participation in another investigational study;
* Inability to follow all study procedures, including attending all site visits, tests and examinations;
* Mental incapacity that precludes adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer I test: to evaluate the performance of "Optrex Double Action soothing and lubricating drops" as soothing and lubricating eye drops for itchy and watery eyes, through the Schirmer I test | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI): to evaluate the performance of "Optrex Double Action soothing and lubricating drops" used to provide relief from eye discomfort associated with itchy and watery eyes, through OSDI | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)
To evaluate the safety and tolerability of "Optrex Double Action soothing and lubricating drops" through Visual Analogue Scale (VAS) - evaluation of symptoms related to dry eye disease (burning, fatigue, discomfort, redness) | End of study visit (EOS/V2 = Day 30 ± 2)
  Visual Analogue Scale:
  Minimum value = 0; Maximum value = 10; Higher scores mean a better outcome.
To evaluate the patient satisfaction through a Rensis Likert 5 points patient satisfaction scale | End of study visit (EOS/V2 = Day 30 ± 2)
  Rensis Likert 5 points patient satisfaction scale Minimum value: Very dissatisfied Maximum value: Vert satisfied Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Policlinico Mater Domini - Università Magna Grecia di Catanzaro, Catanzaro, CZ, Italy